CLINICAL TRIAL: NCT00323401
Title: The Influence of Antenatal Classes on Pregnancy, Birth and Parenthood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital Skejby (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RDM2006
Record Dates: First submitted 2006-05-08; First posted 2006-05-09 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2015-11

CONDITIONS: Pregnancy; Parturition
Keywords: Pregnancy; Parturition; Depression; Randomized; Antenatal classes
MeSH Terms: conditions — Depression | interventions — Prenatal Education; Analgesia; Coping Skills; Lactation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventon (Experimental): Antenatal classes for the parents
  Interventions: Other: Antenatal classes
- Control (No Intervention): No programme are offered

INTERVENTIONS:
Other: Antenatal classes — 3 sessions of 3 hours each
  Other Names: 1. The delivery process, pain relief and coping strategy; 2. Infant care and breastfeeding; 3. The parental role and the relationship
  Arms: Interventon

SUMMARY:
1. To study the influence of antenatal classes for first time parents and their effect ob pregnancy, birth and parenthood.
2. Randomized into two groups (a. 3 courses in midpregnancy and b. no courses)
3. Data on pregnancy, birth and parenthood are collected from register and questionaire

DETAILED DESCRIPTION:
Data collected contain register data and data from questionnaire, which also contains psychometric tests

ELIGIBILITY:
Inclusion Criteria:

Pregnant Over 18 years of age Singleton

Exclusion Criteria:

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1192 (Actual)
Dates: Start 2006-05; Primary Completion 2009-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Arrival for birth | prospective
Birth experience | prospective
Medical interventions during delivery | prospective
Use of birth analgesia | prospective

SECONDARY OUTCOMES:
Length of Birth | prospective
Post partum depression | prospective
Breastfeeding duration and experience | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Jørn Olsen, Professor, Study Chair — University of Aarhus, Department of Epidemiology
Locations (2):
- Denmark (2):
  - University of Aarhus and University Hospital, Skejby, Aarhus
  - Skejby Sygehus, Aarhus

REFERENCES:
- [Derived] Maimburg RD, Vaeth M, Hvidman L, Durr J, Olsen J. Women's worries in first pregnancy: results from a randomised controlled trial. Sex Reprod Healthc. 2013 Dec;4(4):129-31. doi: 10.1016/j.srhc.2013.10.001. Epub 2013 Oct 9. PMID 24216040
- See also: Published results — https://www.ncbi.nlm.nih.gov/pubmed/20536430